CLINICAL TRIAL: NCT03398291
Title: Simultaneous Resection of Pancreatic Cancer and Liver Oligometastasis After Induction Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Chair of Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-1
Record Dates: First submitted 2018-01-01; First posted 2018-01-12 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer; Liver Metastases; Surgery
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Patients continue to receive standard chemotherapy.
  Interventions: Drug: Standard chemotherapy
- Surgical exploration (Experimental): Patients receive surgical exploration and synchronous resection of primary pancreatic cancer and liver oligometastasis will be performed.
  Interventions: Procedure: Synchronous resection of primary pancreatic cancer and liver oligometastasis

INTERVENTIONS:
Procedure: Synchronous resection of primary pancreatic cancer and liver oligometastasis — Patients undergo surgical exploration. If no extensive metastatic sites are found, the synchronous resection of primary pancreatic cancer and liver metastatic sites will be performed. Adjuvant chemotherapy was recommended, and the regimen selection is recommended to be based on the preoperative chemotherapy.
  Arms: Surgical exploration
Drug: Standard chemotherapy — Patients continue to receive standard chemotherapy including folinic acid, fluorouracil, irinotecan and oxaliplatin (FOLFIRINOX), gemcitabine plus nab-paclitaxel, or gemcitabine plus S-1
  Arms: Standard treatment

SUMMARY:
This study is a multi-center phase 3 trial to evaluate a treatment strategy for selecting patients who can benefit from the synchronous resection of primary pancreatic cancer and liver oligometastasis after induction chemotherapy. Half of participants who meet the entry criterion will receive surgical intervention, while the other half will continue to receive standard chemotherapy.

ELIGIBILITY:
Note: This study has two steps. In the first step, patients who meet the criteria for candidates will receive standard first-line chemotherapy for pancreatic cancer. Response Evaluation Criteria in Solid Tumors (RECIST) criteria was employed to measure tumor's response to chemotherapy every two cycles. Until some of them meet the criteria for intervention, they will be randomized and receive relevant interventions.

Inclusion Criteria for candidates:

1. Voluntary participation
2. 18-75 years old
3. Eastern Cooperative Oncology Group (ECOG) 0-1
4. Stage IV pancreatic cancer with no more than 3 liver metastases
5. Histologically confirmed diagnosis of pancreatic cancer
6. No contraindication of chemotherapy

Exclusion Criteria for candidates:

1. Not want to receive chemotherapy or potential operation.
2. Metastases at other sites except for liver
3. With other malignancies
4. Receive chemotherapy, radiotherapy, and interventional therapy before
5. Contraindication of potential operation

Inclusion Criteria for intervention:

1. Primary tumor and liver metastatic sites are both resectable.
2. No new metastatic sites were observed
3. Abnormal serum tumor maker levels decreased by more than 50% after chemotherapy. In the serum tumor makers, carbohydrate antigen 19-9 (CA19-9) was always the first choice for evaluation and it should be below 500U/L after treatment. However, when the baseline CA19-9 was within the normal range, carbohydrate antigen 125 (CA125) and carcinoembryonic antigen (CEA) were the alternative candidate indicators.

Exclusion Criteria for intervention:

1. Contraindication of operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Real overall survival | Up to 2 years
  Including the time of induction chemotherapy

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Not including the time of induction chemotherapy
Life quality score | Up to 2 years, every 2 months
  Quality of life will be measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30
Postoperative morbidity | Up to 90 days after operation
  Including pancreatic fistula, biliary fistula, hemorrhage, wound infection, delayed gastric emptying, reoperation
Postoperative mortality | Up to 90 days after operation
  Patients die from any cause during 90 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Michalski CW, Erkan M, Huser N, Muller MW, Hartel M, Friess H, Kleeff J. Resection of primary pancreatic cancer and liver metastasis: a systematic review. Dig Surg. 2008;25(6):473-80. doi: 10.1159/000184739. Epub 2009 Feb 12. PMID 19212120
- [Background] Cannistra' M, Ruggiero M, Zullo A, Grande R, Nardo B. Surgical resection of synchronous and metachronous metastases from pancreatic adenocarcinoma. Two case reports in the light of recent evidences. Ann Ital Chir. 2015 Dec 29;86(ePub):S2239253X15024160. PMID 26754676
- [Background] Buc E, Orry D, Antomarchi O, Gagniere J, Da Ines D, Pezet D. Resection of pancreatic ductal adenocarcinoma with synchronous distant metastasis: is it worthwhile? World J Surg Oncol. 2014 Nov 18;12:347. doi: 10.1186/1477-7819-12-347. PMID 25407113
- [Background] Zanini N, Lombardi R, Masetti M, Giordano M, Landolfo G, Jovine E. Surgery for isolated liver metastases from pancreatic cancer. Updates Surg. 2015 Mar;67(1):19-25. doi: 10.1007/s13304-015-0283-6. Epub 2015 Feb 22. PMID 25702263
- [Background] Tachezy M, Gebauer F, Janot M, Uhl W, Zerbi A, Montorsi M, Perinel J, Adham M, Dervenis C, Agalianos C, Malleo G, Maggino L, Stein A, Izbicki JR, Bockhorn M. Synchronous resections of hepatic oligometastatic pancreatic cancer: Disputing a principle in a time of safe pancreatic operations in a retrospective multicenter analysis. Surgery. 2016 Jul;160(1):136-144. doi: 10.1016/j.surg.2016.02.019. Epub 2016 Apr 3. PMID 27048934
- [Derived] Wei M, Shi S, Hua J, Xu J, Yu X; Chinese Study Group for Pancreatic Cancer (CSPAC). Simultaneous resection of the primary tumour and liver metastases after conversion chemotherapy versus standard therapy in pancreatic cancer with liver oligometastasis: protocol of a multicentre, prospective, randomised phase III control trial (CSPAC-1). BMJ Open. 2019 Dec 8;9(12):e033452. doi: 10.1136/bmjopen-2019-033452. PMID 31818843